CLINICAL TRIAL: NCT01613651
Title: A Prospective Randomized Trial of Pelvic Drain Placement Versus no Pelvic Drain Placement After Robotic Assisted Laparoscopic Prostatectomy (RALP) in Patients With Prostate Cancer
Brief Title: Robotic Assisted Laparoscopic Prostatectomy With or Without Pelvic Drain Placement in Reducing Adverse Events After Surgery in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11113; NCI-2012-00558 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Perioperative/Postoperative Complications; Prostate Cancer
MeSH Terms: conditions — Postoperative Complications; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (RALP) (Experimental): Patients undergo RALP.
  Interventions: Procedure: robot-assisted laparoscopic surgery; Other: questionnaire administration
- Arm II (RALP and placement of pelvic drain) (Experimental): Patients undergo RALP and placement of pelvic drain.
  Interventions: Procedure: robot-assisted laparoscopic surgery; Other: questionnaire administration; Other: intraoperative complication management/prevention

INTERVENTIONS:
Procedure: robot-assisted laparoscopic surgery — Undergo RALP
Other: questionnaire administration — Ancillary studies
Other: intraoperative complication management/prevention — Undergo placement of pelvic drain
  Arms: Arm II (RALP and placement of pelvic drain)

SUMMARY:
This randomized phase III trial studies robotic assisted laparoscopic prostatectomy (RALP) with pelvic drain placement to see how well it works compared to RALP without pelvic drain replacement in reducing adverse events after surgery in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if eliminating placement of a pelvic drain in patients during robotic assisted laparoscopic prostatectomy (RALP) increases incidence of early postoperative adverse events occurring within 90 days from prostatectomy, compared to patients who have a pelvic drain placed during RALP.

SECONDARY OBJECTIVES:

I. To determine the incidence of early postoperative adverse events in patients with and without a pelvic drain when adjustments to confounders associated with these events are made (confounders: demographic, surgical and pathologic; age, body mass index [BMI], pathologic stage, Gleason sum, extent of lymph node dissection).

II. To report peri-operative and postoperative outcomes, including but not limited to, length of hospital stay, re-admissions, continence, potency and incidence of medical interventions for patients with and without pelvic drain.

III. To compare early postoperative adverse event rates between patients with and without a pelvic drain in patients who had extended pelvic lymph node dissection during RALP.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo RALP.

ARM II: Patients undergo RALP and placement of pelvic drain.

After completion of treatment, patients are followed up at 1 week and then 1, 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male patients diagnosed with prostate cancer and scheduled to undergo RALP at City of Hope National Medical Center
* Written informed consent obtained in accordance with institutional policies approved by the U.S. Department of Health and Human Services
* Patients with prior transurethral resection and other prostate procedures are eligible with the exception of the procedures indicated in the exclusion criteria

Exclusion Criteria:

* Non-compliance
* Prior radiotherapy to the pelvis or prostate
* Prior extensive pelvic surgery such as low anterior reception, abdomino-perineal resection, or proctocolectomy continent stool pouch, or any other extensive abdomino-pelvic surgery that would render the patient high-rick for complications as deemed by the surgeon
* Demonstrated intra-operative anastomotic leakage when irrigated with 120 mL of normal saline at the end of surgery
* Intra-operative injuries (for example: rectal injury)
* Inadequate hemostasis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2012-08-24 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Incidence of early postoperative adverse events according to Common Terminology Criteria for Adverse Events 4.0 (CTCAE 4.0) | Within 90 days from prostatectomy
  The observed rate of adverse events among patients on the two arms of the study will be compared using a one-sided non-inferiority test with the intent to rule out a 10% or greater difference in postoperative adverse event rates.

SECONDARY OUTCOMES:
Incidence of early postoperative adverse events in patients with and without pelvic drain with adjustments applied to confounders associated with these events according to CTCAE 4.0 | Within 90 days post prostatectomy
  Further analysis will be conducted using multivariate logistic regression, to determine whether the odds of early postoperative adverse events are significantly different for patients in different study arms, once they have controlled for confounding prognostic factors, such as age, BMI, pathologic stage, Gleason sum, and lymph node dissection template. Secondary postoperative categorical or continuous endpoints will be examined between arm I and arm II and will be analyzed using the Chi Square T-test, the Mann Whitney test, or the two-sided t-test.
Peri-operative outcomes for patients with and without a pelvic drain, including continence and potency | Up to 12 months
  Survival analysis will be used to determine if there is any significant difference between patients on two arms of the study with respect to time to continence or potency. Secondary postoperative categorical or continuous endpoints will be examined between arm I and arm II and will be analyzed using the Chi Square T-test, the Mann Whitney test, or the two-sided t-test.
Incidence of early postoperative adverse events from prostatectomy in patients with and without a pelvic drain who had an extended pelvic lymph node dissection during RALP according to CTCAE 4.0 | Within 90 days from prostatectomy
  Secondary postoperative categorical or continuous endpoints will be examined between arm I and arm II and will be analyzed using the Chi Square T-test, the Mann Whitney test, or the two-sided t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Yamzon, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States